CLINICAL TRIAL: NCT04645303
Title: Ultrasound-Guided Injection of Hyaluronic Acid Versus Corticosteroid for Treatment of Trigger Finger: Randomized Controlled Study
Brief Title: Injection of Hyaluronic Acid Versus Corticosteroid for Treatment of Trigger Finger
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dubai Health Authority (Other Government)
Responsible Party: Principal Investigator, Sahar Said Khalil, Specialist Senior Registrar- Physical Medicine and Rehabilitation Department- Dubai Hospital- UAE( co-affiliation: Assistant Professor Rheumatology, physical Medicine and rehabilitation- Zagazig University- Egypt), Dubai Health Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSREC-12/2019_03
Record Dates: First submitted 2020-11-04; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Trigger Finger
Keywords: Trigger finger; Hyaluronic Acid; Corticosteroid; Ultrasound-guided injection
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Hyaluronic Acid; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyaluronic acid (Experimental): 1mL of hyaluronic acid (20 mg/2 mL; Hyalgan, Fidia, Abano Terme, Italy) infiltration at A1-Pulley under ultrasound guidance after subcutaneous 2% lidocaine without epinephrine infiltration of the skin overlying the A1-pulley.
  Interventions: Drug: hyaluronic acid (20 mg/2 mL)
- Triamcinolone acetonide (Active Comparator): 1 mL of Triamcinolone acetonide 10mg/ml infiltration at A1-Pulley under ultrasound guidance after subcutaneous 2% lidocaine without epinephrine infiltration of the skin overlying the A1 pulley.
  Interventions: Drug: Triamcinolone acetonide 10mg/ml

INTERVENTIONS:
Drug: hyaluronic acid (20 mg/2 mL) — A1-Pulley infiltration for trigger finger
  Other Names: Hyalgan 20 mg in 2 ML Prefilled Syringe
  Arms: Hyaluronic acid
Drug: Triamcinolone acetonide 10mg/ml — A1-Pulley infiltration for trigger finger
  Other Names: Kenalog 10 mg/ml
  Arms: Triamcinolone acetonide

SUMMARY:
The aim of the study is to compare the therapeutic effects of hyaluronic acid versus steroid injections in treating trigger fingers using ultrasound guidance

DETAILED DESCRIPTION:
A prospective randomized controlled study designed to compare the outcomes of injecting patients with trigger finger with hyaluronic acid versus corticosteroid under ultrasound guidance

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* Patients with a clinical diagnosis of trigger finger grade 1-3 on the Quinnell grading scale and confirmed diagnosis by ultrasound.

Exclusion Criteria:

* Quinnell's classification grade IV (contracture)
* Prior injection within 6 months
* Prior operation of the affected finger
* Presence of any contracture in the proximal interphalangeal or metacarpophalangeal joint, and
* History of diabetes, hypothyroidism, and
* Rheumatic or connective tissue disease
* Allergy to triamcinolone or hyaluronic acid
* Pregnancy
* Secondary triggering e.g. Trauma, infection
* Trigger finger symptoms duration >6 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-04-05 (Estimated); Study Completion 2021-06-04 (Estimated)

PRIMARY OUTCOMES:
Change in Quinnell trigger finger grading system: | 1 and 3 months post-injection
  Change in Quinnell grading overtime within 3 months after injection. Trigger fingers are rated as follows: Grade 0: normal finger movements, Grade 1: uneven finger movements, Grade 2: actively correctable triggering, Grade 3: passively correctable triggering, and Grade 4: locked digit.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) of pain | 1 and 3 months post-injection
  Change in pain Visual analogue scale will be recorded. The patient marks on the 100 mm in length line the point that he/she feels to represent his/her perception of pain at the current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks ( a higher score indicates greater pain intensity). Categorization of none, mild, moderate and severe pain will be also used (none = 0, mild = 1-4, moderate = 5-6, and severe = 7-10).
Frequency of tender trigger nodules | 1 and 3 months post-injection
  Identifying the presence of tender nodules at A1-pulley of the affected finger by palpation
The Quick Disability of the Arm, Shoulder and Hand score | 1 and 3 months post-injection
  Patients will be asked to fill a questionnaire form. It is an 11-item form that assesses the upper limb function on a scale of 1-5, with scores ranging from 11 to 55, with the higher scores representing more disability and worse upper limb function.
Changes in Grip strength | 1 and 3 months post-injection
  Measured by the dynamometer strength test (Jamar grip dynamometer)
Patient satisfaction with therapy | 1 and 3 months post-injection
  Participating patients will be asked to classify their result into 1 of 4 categories: (1) complete resolution of symptoms, (2) improved result, but incomplete resolution of symptoms, not warranting further treatment, (3) partial response, but unsatisfactory, warranting further treatment, and (4) no response.
Ultrasound evaluation of A1-Pulley | 1 and 3 months post-injection
  Detailed ultrasonography evaluation of A1-Pulley. Comparing the A1-Pulley ultrasonographic parameters over 3 months after injection (at the follow-up appointment)

CONTACTS AND LOCATIONS:
Overall Officials: Sahar S Khalil, SSR, Principal Investigator — Specialist Senior Registrar- Physical Medicine and rehabilitation Department- Dubai hospital; Mohamed M Abdulla, Consultant, Study Chair — Consultant and Head of Physical Medicine and rehabilitation Department- Dubai hospital
Locations (1):
- Dubai Hospital- Dubai Health Authority, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu DH, Tsai MW, Lin SH, Chou CL, Chiu JW, Chiang CC, Kao CL. Ultrasound-Guided Hyaluronic Acid Injections for Trigger Finger: A Double-Blinded, Randomized Controlled Trial. Arch Phys Med Rehabil. 2015 Dec;96(12):2120-7. doi: 10.1016/j.apmr.2015.08.421. Epub 2015 Sep 1. PMID 26340807
- [Background] Callegari L, Spano E, Bini A, Valli F, Genovese E, Fugazzola C. Ultrasound-guided injection of a corticosteroid and hyaluronic acid: a potential new approach to the treatment of trigger finger. Drugs R D. 2011;11(2):137-45. doi: 10.2165/11591220-000000000-00000. PMID 21545190
- [Background] Abate M, Schiavone C, Salini V. The use of hyaluronic acid after tendon surgery and in tendinopathies. Biomed Res Int. 2014;2014:783632. doi: 10.1155/2014/783632. Epub 2014 May 8. PMID 24895610